CLINICAL TRIAL: NCT03104608
Title: Automatic Self Transcending Meditation (ASTM) Plus Treatment As Usual (TAU) Versus TAU Alone in Patients With Severe Age Related Macular Degeneration (AMD), a Single Blind Randomized Controlled Longitudinal Study
Brief Title: Automatic Self Transcending Meditation (ASTM) for Patients With Severe Age Related Macular Degeneration (AMD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Monali Malvankar, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10016731
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Age-related Macular Degeneration; Low Vision
MeSH Terms: conditions — Macular Degeneration; Vision, Low | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Self Transcending Meditation (Active Comparator): Participants in the ASTM group will undergo training in groups of 10 by certified teachers. Further, the following self-rated scales will be administered by a trained rater at the fourth ASTM session (week 0) as well as at weeks 4, 8, 12, and 24: Time Trade-off (TTO), Visual Function Questionnaire (VFQ-25), the Patient Health Questionnaire (PHQ-9), and Generalized Anxiety Disorder (GAD-7).
  Interventions: Other: Automatic Self Transcending Meditation
- Treatment as Usual (Placebo Comparator): Participants will continue to receive their treatment as usual. The following self-rated scales will be administered by a trained rater at weeks 0, 4, 8, 12 and 24: TTO, VFQ-25, PHQ-9, and GAD-7.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Automatic Self Transcending Meditation — Automatic Self Transcending Meditation is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness. Research suggests that ASTM is easier to learn and to teach in comparison to other meditation techniques. Further, studies have shown that ASTM confers large effect sizes as an anti-depressant.
  Arms: Automatic Self Transcending Meditation
Other: Treatment as Usual — Participants randomized to Treatment as Usual (TAU)) will continue to receive their treatment as usual.
  Arms: Treatment as Usual

SUMMARY:
Age-related macular degeneration (AMD) is a condition affecting 20 to 25 million people worldwide. Symptoms of AMD includes difficulty in reading, recognizing faces and completing house work which may result in increased disability which in turn increase symptoms of depression and anxiety. Depression and anxiety could also be worsened by social isolation caused by AMD. Further, AMD causes high levels of emotional distress and reduced quality of life (QoL). Automatic Self Transcending Meditation (ASTM) - a standardized category of meditation - may help reduce stress, depression, anxiety, and may enhance QoL. Automatic Self Transcending Meditation (ASTM) is a class of meditation that helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. It utilizes a specific sound value (mantra) to draw attention inward and permit the mind to experience a restful but alert state of consciousness. In the proposed research, the effects of ASTM on health related quality of Life (HRQoL), depression and anxiety in low-vision AMD patients will be studied. A single-center, single-blind longitudinal randomized controlled trial (RCT) will be conducted in London, ON. Patients with AMD (n = 140, 70 in each arm) will be randomized to ASTM plus treatment as usual (TAU) or TAU alone (control) arm. Data on routinely measured ophthalmic clinical variables, HRQoL, depression, and anxiety will be collected from both the arms. Statistical analysis will be conducted using STATA 15.0 to evaluate the effects of ASTM plus TAU compared to TAU alone on HRQoL, depression, and anxiety. Further, for each group - ASTM plus TAU and TAU alone - the investigators develop an association between HRQoL, depression, and anxiety with routinely measured clinical variables using mathematical models.

DETAILED DESCRIPTION:
OBJECTIVE: The investigators key objective is to study the effects of ASTM on HRQoL, depression, and anxiety in AMD patients. The second objective is to determine if there is an association between HRQoL, depression, and anxiety with routinely measured clinical variables. A mathematical model to compute HRQoL, depression, and anxiety from ophthalmic clinical variables will be developed in ASTM plus TAU as well as TAU alone group.

Study Design: The investigators plan to conduct a single-center, single blind longitudinal randomized controlled trial (RCT). Research participants will be 140 men and women (70 in each group).

Study Recruitment: Potential participants with severe AMD above 50 years of age will be screened - from the office practice of Dr. Mao as per inclusion and exclusion criteria at the Ivey Eye Institute, London, ON.

An ophthalmic examination - offered as a routine care - for each potential participant (i.e., measuring best-corrected Snellen visual acuity and pinhole acuities) will be conducted. Snellen acuity will be converted to LogMAR according to visual angle subtended by letters such as 20/20 = 0.0, 20/40 = 0.3, 20/50 = 0.3978. A value above 20/200 = 1.0 will be assigned to counting fingers, hand motions, and light perception. No light perception will receive a value of 0.0.

Questionnaire: Patients will undergo a standardized interview performed by a trained interviewer to measure HRQoL using the time trade-off method (TTO) in which potential participants will be asked couple of questions about their quality of life such as 1) how long participant expect to live? and 2) how many of those remaining years of life, if any, participant would be willing to trade in return for a treatment permitting to their current vision in each eye to be transformed to permanent perfect vision (20/20) bilaterally?. During the first office visit (screening visit), in the interview, patients will be asked demographic questions including age, gender, and associated medical conditions, such as concurrent ocular conditions, ocular disease other than AMD, previous ocular surgery, intraoperative complications, preoperative ocular pathology, chronic pain, general diseases that could affect the immune system, and actual infection. In addition, patients will be asked about co-morbidities such as, whether they have high blood pressure, diabetes, arthritis, heart condition, stroke, and other non-ocular medical conditions. Further, the following self-rated scales will be administered at the first office visit: TTO, Visual Function Questionnaire (VFQ-25), the Patient Health Questionnaire (PHQ-9), and Generalized Anxiety Disorder (GAD-7).

Randomization: Participants will be randomized to ASTM + TAU or TAU alone equally (1:1) using computer generated randomization numbers available at random.org. Concealment of randomization will be ensured by independent staff performing randomization using a third party web-based provider (http://www.sealedenvelope.com/). Computerized randomization will occur from the Ivey Eye Institute, St. Joseph's Hospital, London, ON. A telephone number will be available for study concerns/queries. Pre-randomized information will be stored using unique de-identifiers and downloaded on a secure database. Outcome assessors and investigators will be blinded to treatment.

Trial Interventions/Treatment Arms: 1) Automatic Self-Transcending meditation (ASTM): Following the initial measurements (common to both ASTM and control group), participants in the ASTM group will undergo ASTM training in groups of 10 by certified teachers under the supervision of one of the study collaborator at a room in St. Joseph's Hospital, London, ON. This involves participating in four, 90-120 minute sessions each of four consecutive days. This will be followed by weekly 60 minute follow up sessions for 4 weeks, biweekly sessions for weeks 5-12 weeks and monthly follow-up session for 13-24 weeks. Participants will be required to attend 75% of weekly, bi-weekly, monthly follow-up sessions. In addition, participants will be asked to practice ASTM at home for 20 minutes twice daily over the study period (24 weeks). Participants will be asked to log practice frequency and any other noteworthy observations in the log sheet provided to them. Further, the following self-rated scales will be administered by a trained rater at the fourth ASTM session (week 0) as well as at weeks 4, 8, 12, and 24: TTO, VFQ-25, PHQ-9, and GAD-7 Questionnaire. 2) Control Intervention: Participants randomized to control arm (Treatment as Usual (TAU)) will continue to receive their treatment as usual. They will follow assessment and study procedures as listed below. The following self-rated scales will be administered by a trained rater at weeks 0, 4, 8, 12 and 24: TTO, VFQ-25, PHQ-9, and GAD-7. No study procedures will be applied or any other information collected during this period. All medication types will be permitted in this study. Any dosage modifications will be recorded. The investigators anticipate to recruit participants at a rate of at least 10 participants/week over a period of 7 weeks allowing attainment of sample size of n=140. There is no obligation for the participants to take part in the study; all participation is voluntary.

Sample Size: Health Related Quality of Life (HRQoL) was chosen as the main covariate of interest. Based on literature, sample size computations were performed, for alpha = 0.05, 80% power, 1.0 as mean HRQoL of ASTM + TAU group and 0.5 as mean HRQoL of TAU alone group, the investigators estimated the sample size using a two-sample means test assuming equal variances to be 128, 64 per group. A sample size of 140 (70 in each arm) to account for attrition and loss of data from follow ups at an average of 10-15% will be recruited. Such a moderate attrition rate is expected based on previously published studies as well as our own ongoing studies.

Data Analysis:

Dependent variable: A dependent variable is created based on the HRQoL, an interval scale variable taking values between 0.0 and 1.0.

Independent variables: Visual acuity in a better-seeing eye, patients' demographic characteristics, including age, gender, and associated medical conditions are the independent variables. Patients' demographic characteristics, including age, are considered as continuous variables. Gender is categorized as male and female and associated medical conditions are categorized as "current medical conditions," which includes concurrent ocular conditions; "other diseases," which includes ocular diseases other than AMD, chronic pain, general diseases that could affect the immune system, and actual infection; and "medical history," which includes previous ocular surgery, preoperative ocular pathology, and intraoperative complications.

Data Grouping: Based on BCVA, study participants will be grouped to visual acuity in better seeing eye (group 1, 20/20 to 20/50; group 2, 20/60 to 20/100; group 3, 20/200 to no light perception). Better seeing will be used since a correlation has been shown between utility score and better seeing eye. These 3 groups were chosen since group 1 represents legal driving vision in Canada, group 2 represents moderate visual acuity loss, and group 3 represents legal blindness.

Analysis: As has been done in many other studies, HRQoL will be calculated by dividing the number of years a patient is willing to trade in return for improved quality of life by the estimated numbers of years of remaining life subtracted by 1.0 as given below: HRQoL(U)=1-(number of years a patient is willing to trade in return for improved quality of life)/(estimated number of years of remaining life). Mean, standard deviation, and 95% confidence interval for continuous variables such as utility value, will be calculated. For categorical variables, visual acuity in the better-seeing eye, gender, and associated medical conditions, proportions will be calculated. The chi-square test statistic for independence will be used to compare unwillingness to trade time in TTO. The unpaired, two-tailed Student t-test will be used to evaluate the effect of visual acuity in the better eye in four groups and gender on mean of TTO utility values. Non-response issues: Non-respondent patients' characteristics will be compared with respondent patients,' and if they do not appear to be statistically significantly different, then these results will be generalized to the sample and population.

Data will be analyzed using STATA Software. The unit of analysis is the HRQoL. Univariate and bivariate analysis will be performed for each independent variable against the dependent variable to elicit the impact of each factor on the pattern of HRQoL without adjusting for the effect of other variables. Models will be deemed statistically significant if they are associated with a significant F value (p < 0.01) and if they explain over 15% variability of the dependent variable. Only those independent variables that are statistically significantly associated with the HRQoL (p < 0.05) will be used for model construction. Since the dependent variable is continuous, the investigators plan to use a non-linear regression model to assess the effect of each independent variable on the dependent variable, while controlling for the confounders. Multicollinearity, high correlation between independent variables, and interaction effects will be evaluated for the model.

Validation Analysis: Validation will be performed on the developed regression model. The collected data will be divided into two portions: one portion, called the "main data," will contain 80% of the samples of the total collected utility values and its associated data; the other portion, called the "test data," will contain the remaining 20%. Validation will be done using test data but having the same coefficient values as the main data in order to calculate the percentage of correct cases. Similar regression analysis as described above will be performed for each dependent variable: vision related quality of life measured by VFQ-25, depression score measured by PHQ-9, and anxiety score measured by GAD-7.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years of age,
* have severe AMD
* deemed competent such as no language issues or communication barriers, no self-reported or physician diagnosed mental health disorder besides having depressive and anxiety symptoms
* have sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 30 minutes
* willing and able to attend 4 initial ASTM training sessions and at least 75% of weekly, bi-weekly and monthly follow up sessions
* willing to dedicate 20 minutes twice per day to ASTM practice at their own home.

Exclusion Criteria:

* actively suicidal as per self-report (scoring 2 or more on item 9 of the Patient Health Questionnaire (PHQ-9) or on assessment by the physician
* they are currently participating in other similar studies
* currently practicing any type of formal meditation regularly
* unable or unwilling to answer survey questions.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life (HRQoL) | Change from baseline up to 24 weeks
  HRQoL is measured using the time trade-off method (TTO) in which potential participants will be asked couple of questions about their quality of life such as 1) how long participant expect to live? and 2) how many of those remaining years of life, if any, participant would be willing to trade in return for a treatment permitting your current vision in each eye to be transformed to permanent perfect vision (20/20) bilaterally?.

SECONDARY OUTCOMES:
Change in Vision Score | Change from baseline up to 24 weeks
  Visual Function Questionnaire (VFQ-25) will be used to measure vision score
Change in Depression score | Change from baseline up to 24 weeks
  Patient Health Questionnaire (PHQ-9) will be used to measure depression score
Change in Anxiety score | Change from baseline up to 24 weeks
  Generalized Anxiety Disorder (GAD-7) will be used to measure anxiety score

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers. The investigators have the expertise to perform statistical analysis so do not need outside help.

REFERENCES:
- [Result] Hamade N, Hodge WG, Rakibuz-Zaman M, Malvankar-Mehta MS. The Effects of Low-Vision Rehabilitation on Reading Speed and Depression in Age Related Macular Degeneration: A Meta-Analysis. PLoS One. 2016 Jul 14;11(7):e0159254. doi: 10.1371/journal.pone.0159254. eCollection 2016. PMID 27414030